CLINICAL TRIAL: NCT00115310
Title: A Randomized, Double-Blind, Controlled Study of NGX-4010 for the Treatment of Postherpetic Neuralgia
Brief Title: Study of NGX-4010 for the Treatment of Postherpetic Neuralgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NeurogesX (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C116
Record Dates: First submitted 2005-06-21; First posted 2005-06-22 (Estimated); Last update posted 2008-03-06 (Estimated); Status verified 2008-03

CONDITIONS: Peripheral Nervous System Diseases; Pain; Neuralgia; Herpes Zoster; Shingles
Keywords: dermal assessment; pain measurement; diary; PHN; shingles; neuropathy; analgesics; capsaicin; postherpetic neuralgia
MeSH Terms: conditions — Peripheral Nervous System Diseases; Pain; Neuralgia; Herpes Zoster; Neuralgia, Postherpetic | interventions — Capsaicin

INTERVENTIONS:
Drug: NGX-4010

SUMMARY:
The purpose of the study is to assess the efficacy and safety of NGX-4010 applied for 60 minutes for the treatment of postherpetic neuralgia (PHN).

DETAILED DESCRIPTION:
This study is a 12-week randomized, double-blind, controlled multi-center evaluation of the efficacy, safety and tolerability of NGX-4010 for the treatment of PHN. Eligible subjects will have moderate to severe pain from PHN, with average NPRS scores during screening of 3 to 9 (inclusive). Painful areas of up to 1000 square centimeters will be treated during a single treatment administration in this study. Subjects will be randomly assigned to receive active NGX-4010 patches or low-concentration control patches that are identical in appearance, according to a 1:1 allocation scheme.

Subjects may be on stable chronic oral pain medication regimens, but currently will not be using any topical pain medications on the affected areas. NPRS scores for the average pain in the past 24 hours will be recorded daily in the evening, beginning on the day of the Screening Visit (usually on Day -14). Subjects will continue to record NPRS scores in a take-home diary from the evening on the day of treatment through the evening before the Termination Visit at Week 12. Subjects will return for interim follow-up visits at Weeks 4 and 8 following study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PHN, with at least 6 months of pain since shingles vesicle crusting
* Average NPRS scores for PHN-associated pain during screening period of 3 to 9
* Intact, unbroken skin over the painful area(s) to be treated
* If taking chronic pain medications, be on a stable (not PRN) regimen for at least 21 days prior to Study Patch Application Visit (Day 0) and willing to maintain medications at same stable dose(s) and schedule throughout study
* Female subjects with child-bearing potential must have a negative serum beta human chorionic gonadotropin (hCG) pregnancy test, within 7 days of Study Patch Application Visit
* All subjects must be willing to use effective methods of birth control and/or refrain from participating in a conception process during the study (or, in the event of early termination from the study, for 30 days following experimental drug exposure)
* Be willing and able to comply with protocol requirements for the duration of study participation.
* Subjects must sign an informed consent form for this study approved by the Investigator's Institutional Review Board/Independent Ethics Committee (IRB/IEC).

Exclusion Criteria:

* Concomitant opioid medication, unless orally or transdermally administered and not exceeding a total daily dose of morphine 60 mg/day, or equivalent. Parenteral opioid use is excluded, regardless of dose.
* Unavailability of an effective rescue medication strategy for the subject, such as unwillingness to use opioid analgesics during study treatment, or high tolerance to opioids precluding the ability to relieve treatment-associated discomfort, as judged by Investigator.
* Active substance abuse or history of chronic substance abuse within the past year, or prior chronic substance abuse (including alcoholism) judged likely to recur during the study period by Investigator.
* Recent use (within 21 days preceding the Study Patch Application Visit [Day 0]) of any topically applied pain medication, such as non-steroidal anti-inflammatory drugs, menthol, methyl salicylate, local anesthetics including Lidoderm (lidocaine patch 5%), steroids or capsaicin products on the painful areas.
* Participation in a previous NeurogesX clinical trial in which subject received NGX-4010 (either blinded or open-label study treatment).
* Current use of any investigational agent, or Class 1 anti-arrhythmic drugs (such as tocainide and mexiletine).
* Diabetes mellitus, unless well-controlled as evidenced by an HbA1c level less than or equal to 9%.
* Hypertension, unless adequately controlled by medication.
* Significant pain of an etiology other than PHN. Subjects must not have significant ongoing pain from other cause(s) that may interfere with judging PHN-related pain.
* Painful PHN areas located only on the face, above the hairline of the scalp, and/or in proximity to mucous membranes.
* Any implanted medical device (spinal cord stimulator, intrathecal pump or peripheral nerve stimulator) for the treatment of neuropathic pain.
* Hypersensitivity to capsaicin (i.e., chili peppers or OTC capsaicin products), local anesthetics, oxycodone hydrochloride, hydrocodone bitartrate or adhesives.
* Significant ongoing or untreated abnormalities in cardiac, renal, hepatic, or pulmonary function that may interfere either with the ability to complete the study or the evaluation of adverse events.
* Recent history of a significant medical-surgical intervention in the judgment of the Investigator.
* Evidence of cognitive impairment including dementia that may interfere with subject's ability to complete daily pain diaries requiring subject's recall of average PHN pain level in the past 24 hours.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2005-06; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in "average pain for the past 24 hours" Numeric Pain Rating Scale (NPRS) score (i.e., average of scores during Weeks 2 to 8, compared to baseline) in the active group compared to the control group

SECONDARY OUTCOMES:
Percent change from baseline in "average pain for the past 24 hours" NPRS score (i.e., average of scores during Weeks 2 to 4 and 2 to 12, respectively, compared to baseline) in the active group compared to the control group
Proportion of subjects reaching 30% and 50% decrease, respectively, from baseline in "average pain for the past 24 hours" NPRS scores on average during Weeks 2 to 8
Proportion of subjects reaching 30% and 50% decrease, respectively, from baseline in "average pain for the past 24 hours" NPRS scores on average during Weeks 2 to 4 and 2 to 12, respectively
Median onset and mean duration of efficacy in days in the active group
Proportion of subjects with significant changes in concomitant pain medication usage during Weeks 2 to 8, compared to baseline
Brief Pain Inventory (BPI)
Short-Form McGill Pain Questionnaire (SF-MPQ)
Subject Global Impression of Change (PGIC)
Self-Assessment of Treatment (SAT)
Short-Form 36v2 Health Survey (SF-36v2™)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Tobias, MD, Study Director — NeurogesX

REFERENCES:
- [Derived] Backonja M, Wallace MS, Blonsky ER, Cutler BJ, Malan P Jr, Rauck R, Tobias J; NGX-4010 C116 Study Group. NGX-4010, a high-concentration capsaicin patch, for the treatment of postherpetic neuralgia: a randomised, double-blind study. Lancet Neurol. 2008 Dec;7(12):1106-12. doi: 10.1016/S1474-4422(08)70228-X. Epub 2008 Oct 30. PMID 18977178